CLINICAL TRIAL: NCT07244562
Title: Effects of Cognitive Training and Exercise on Cognitive Function in Older Women: the INCOGNITO Randomized Clinical Trial
Brief Title: Effects of Physical Exercise and Cognitive Training on Quality of Life in Older Women
Acronym: INCOGNITO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Fabio Manfredini, Full Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 417/2025/Sper/UniFe
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Elderly; Older Adults, Aging Brain
MeSH Terms: interventions — Exercise; Dosage Forms; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1 - Exercise plus cognitive training (Experimental): In addition to the exercise program, participants will be given a series of cognitive exercises aimed at improving prospective memory through the performance of certain oral tasks, administered by a member of the research team. All cognitive exercises will be adapted to the cognitive abilities of the participants
  Interventions: Behavioral: Exercise plus cognitive training
- Experimental 2 - Exercise plus cognitive stimulus (Experimental): In addition to the exercise program, people randomised into this group will receive a short video lasting less than 10 minutes on their smartphone or tablet before the exercise session (or at home). At the end of the video, they will be asked to complete a 10-question questionnaire (also delivered via smartphone or tablet) with True or False answer options
  Interventions: Behavioral: Exercise plus cognitive stimulus at home
- Active comparator - Exercise only (Active Comparator): The exercise program (equal for all the study groups with the exercise intervention) includes 75-minute training sessions twice a week, for a total of 24 training sessions over 12 weeks. Each training session will be divided into a warm-up, training phase and cool-down, and will include aerobic exercises, resistance training, balance exercises, mobility exercises and stretching.
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Control group (No Intervention): The subjects included in this group will not receive any specific treatment. They will receive advice on how to stay active at home and will undergo scheduled assessments.

INTERVENTIONS:
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — The exercise program includes 75-minute training sessions twice a week, for a total of 24 training sessions over 12 weeks. Each training session will be divided into a warm-up, training phase and cool-down, and will include aerobic exercises, resistance training, balance exercises, mobility exercises and stretching.
  Arms: Active comparator - Exercise only
Behavioral: Exercise plus cognitive training — In addition to the exercise program, participants will be given a series of cognitive exercises aimed at improving prospective memory through the performance of certain oral tasks, administered by a member of the research team. All cognitive exercises will be adapted to the cognitive abilities of the participants.
  Arms: Experimental 1 - Exercise plus cognitive training
Behavioral: Exercise plus cognitive stimulus at home — In addition to the exercise program, participants will receive a short video lasting less than 10 minutes on their smartphone or tablet before the exercise session (or at home). At the end of the video, they will be asked to complete a 10-question questionnaire (also delivered via smartphone or tablet) with True or False answer options.
  Arms: Experimental 2 - Exercise plus cognitive stimulus

SUMMARY:
Ageing exposes people to a progressive loss of cognitive and functional abilities, especially in women. The aim of the study is to investigate the effectiveness of different types of intervention, based on physical exercise and/or cognitive stimulation or training, on quality of life, cognition and mobility, on a population of older women.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 60 years
* Provision of the informed consent form

Exclusion Criteria:

* Absolute contraindications to physical exercise (e.g. Nyha class iv heart failure, unstable angina, etc.)
* Pregnancy
* Severe cognitive impairment, defined as a MoCa score ≤ 12
* Severe visual impairment or blindness

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Executive function and processing speed by the Trail Making Test (TMT) | Baseline; end of the program (3-month); Follow-up (6-month)
  TMT is neuropsychological test that assesses a person's cognitive function, specifically focusing on visual attention, processing speed, and executive function. The test consists of two parts, the score is based on the time it takes to complete each part, with shorter times indicating better performance.

SECONDARY OUTCOMES:
Quality of life by the Quality of Life in Alzheimer's Disease (QOL-AD) questionnaire | Baseline; end of the program (3-month); Follow-up (6-month)
  QOL-AD consists of 13 questions covering various aspects of daily life, such as physical health, energy, mood, relationships and the ability to enjoy enjoyable activities. The combined scores of the patient and caregiver provide a more comprehensive and accurate picture of the person's overall well-being. The scale has a score ranging from 13 (lowest quality of life) to 52 (highest quality of life).
  This measure will be collected in people with MCI only
Quality of life assessed by the short-form 36 (SF-36) questionnaire | Baseline; end of the program (3-month); Follow-up (6-month)
  This is a generic questionnaire that contains 36 questions referring to 8 specific domains related to patient health over the previous 4 weeks. For each specific domain, the score ranges from 0 (lowest quality of life) to 100 (highest quality of life).
Cognition assessed by the Montreal Cognitive Assessment (MoCA) | Baseline; end of the program (3-month); Follow-up (6-month)
  MoCA is a 30-point test evaluates cognitive function. Its primary purpose is to detect mild cognitive impairment (MCI). The score goes from 0 (maximal cognitive deficit) to 30 (normal cognitive function).
Walking endurance assessed by the 6-Minute Walking Test (6MWT) | Baseline; end of the program (3-month); Follow-up (6-month)
  The patients will be instructed to walk back and forth on a 20-meter corridor aiming at covering as much distance as possible. The total distance covered (6MWD) will be measured in meters
Physical performance assessed using the Short Physical Performance Battery (SPPB) | Baseline; end of the program (3-month); Follow-up (6-month)
  It is a specific assessment for the elderly population, consisting of three functional tests that measure postural stability, the ability to walk safely, and lower limb muscle strength. The scale goes from 0 (lowest functional ability) to 12 (highest functional ability).
Manual grip strength using the Handgrip Test (HT). | Baseline; end of the program (3-month); Follow-up (6-month)
  The test is performed using a dynamometer: the subject grabs the handle of the device with maximum strength, and the maximum value of force expressed in kilograms is recorded.
Sleep quality and related disorders through the Pittsburgh Sleep Quality Index (PSQI) | Baseline; end of the program (3-month); Follow-up (6-month)
  It refers to the last 30 days and analyses seven components. The total score ranges from 0 to 21. A score above 5 indicates poor sleep quality.
Frontal and prefrontal cerebral perfusion using near-infrared spectroscopy (fNIRS). | Baseline; end of the program (3-month); Follow-up (6-month)
  Changes in brain metabolism will be assessed using NIRS with a system consisting of 16 sources and 16 detectors emitting two wavelengths of light in the near infrared range. Recording using the non-invasive fNIRS method will take place during the TMT.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Manfredini, MD, PhD, Study Chair — Università degli Studi di Ferrara
Locations (1):
- Esercizio Vita, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided